CLINICAL TRIAL: NCT04976296
Title: Dynamic Molecular Residual Disease Detection in Stage I-IIIA Non-Small Cell Lung Cancer After Radical Resection
Brief Title: MRD Monitoring in Lung Cancer After Resection
Status: Recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Xue-Ning Yang, Principal Investigator, Guangdong Provincial People's Hospital
Other Study IDs: NOTICE study
Record Dates: First submitted 2021-07-19; First posted 2021-07-26 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Lung Cancer
Keywords: Molecular residual disease; Circulating tumor DNA; Disease relapse; Predictive value
MeSH Terms: conditions — Lung Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma cell free DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stage I-IIIA NSCLC patients after complete resection: For stage I-IIIA NSCLC patients who underwent complete resection.
  Interventions: Diagnostic Test: MRD detection

INTERVENTIONS:
Diagnostic Test: MRD detection — The Geneplus OncoMRD lung assay is used to detect the MRD status.
  Other Names: Geneplus OncoMRD lung assay

SUMMARY:
The conception of molecular residual disease (MRD) extending from hematologic tumor to solid tumors. Evidences supporting MRD evaluation for lung cancer by liquid biopsy has gradually accumulated, especially circulating tumor DNA (ctDNA). In this observational study, the investigators prospectively enroll stage I-IIIA non-small cell lung cancer (NSCLC) patients who underwent complete resection. Preoperative blood sample, tumor tissue and dynamic postoperative blood samples are collected continuously for MRD detection. This study aim to explore the prognostic value of MRD for stage I-IIIA NSCLC patients after complete resection.

DETAILED DESCRIPTION:
There will be a rapid surge in research about molecular residual disease (MRD) for solid cancer in the near future. However, MRD differed significantly between tumor types and between contexts; there continues to be a considerable lack of awareness and knowledge about using MRD in lung cancer. Hence, this study aims to investigate the value of MRD in NSCLC patients who underwent complete resection. Preoperative blood sample (20ml), tumor tissue and dynamic postoperative blood samples (20ml) are collected continuously for MRD detection. The follow-up was performed once every 3 to 6 months. The primary objective of this study is to assess the prognostic value of MRD for stage I-IIIA NSCLC patients after complete resection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically confirmed NSCLC (WHO 2015 classification) with resectable (stage I-IIIA) disease.
* Complete resection
* Age ≥18 years at the time of screening
* Capable of giving signed informed consent

Exclusion Criteria:

* Mixed small cell and NSCLC histology
* Rx, R1 or R2 resection
* History of other malignant tumors within 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The pathological diagnosis confirmed stage I-IIIA NSCLC patients who underwent complete resection. No history of other malignant tumors within 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The prognostic value of MRD | 5 year
  The survival difference between MRD positive and MRD negative patients.

SECONDARY OUTCOMES:
The predictive value of MRD | 5 year
  The separative value adjuvant chemotherapy or target therapy in MRD positive population and MRD negative population.
The lead time of MRD | 5 year
  The median lead time of detectable MRD before regular imaging finding.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Lung Cancer Institute & Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
The IPD could be shared after seeking consent from the corresponding investigator.

REFERENCES:
- [Background] Pantel K, Alix-Panabieres C. Liquid biopsy and minimal residual disease - latest advances and implications for cure. Nat Rev Clin Oncol. 2019 Jul;16(7):409-424. doi: 10.1038/s41571-019-0187-3. PMID 30796368
- [Background] Abbosh C, Birkbak NJ, Swanton C. Early stage NSCLC - challenges to implementing ctDNA-based screening and MRD detection. Nat Rev Clin Oncol. 2018 Sep;15(9):577-586. doi: 10.1038/s41571-018-0058-3. PMID 29968853
- [Background] Chaudhuri AA, Chabon JJ, Lovejoy AF, Newman AM, Stehr H, Azad TD, Khodadoust MS, Esfahani MS, Liu CL, Zhou L, Scherer F, Kurtz DM, Say C, Carter JN, Merriott DJ, Dudley JC, Binkley MS, Modlin L, Padda SK, Gensheimer MF, West RB, Shrager JB, Neal JW, Wakelee HA, Loo BW Jr, Alizadeh AA, Diehn M. Early Detection of Molecular Residual Disease in Localized Lung Cancer by Circulating Tumor DNA Profiling. Cancer Discov. 2017 Dec;7(12):1394-1403. doi: 10.1158/2159-8290.CD-17-0716. Epub 2017 Sep 24. PMID 28899864